CLINICAL TRIAL: NCT07243795
Title: Impact of Preoperative Ejaculation or Abstinence on Seminal Vesicle Size and Intraoperative Dissection Parameters During Radical Prostatectomy: A Randomized Controlled Trial
Brief Title: Ejaculatory Behavior and Seminal Vesicle Size During Radical Prostatectomy
Acronym: PreRP-EJAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 202507191RINA
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer Patients Undergoing Radical Prostatectomy
Keywords: Prostate Cancer; Radical Prostatectomy; Seminal Vesicle; Ejaculation; Abstinence; Surgical Dissection
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to either a recent ejaculation group or an abstinence group before radical prostatectomy.
Who Masked: Outcomes Assessor
Masking Description: The operating surgeon was masked to the participant's group assignment. Group allocation was concealed until after surgery. Neither the participant nor the research investigator performing TRUS was masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recent Ejaculation Group (Experimental): Participants in this group will be instructed to have at least one ejaculation within 36 hours before surgery. Under anesthesia, they will undergo transrectal ultrasound (TRUS) to measure seminal vesicle volume prior to radical prostatectomy. Intraoperative dissection time, difficulty, and visual clarity will also be recorded.
  Interventions: Behavioral: Recent Ejaculation
- Abstinence Group (Active Comparator): Participants in this group will be instructed to abstain from ejaculation for at least 72 hours before surgery. Under anesthesia, they will undergo transrectal ultrasound (TRUS) to measure seminal vesicle volume prior to radical prostatectomy. Intraoperative dissection time, difficulty, and visual clarity will also be recorded.
  Interventions: Behavioral: Preoperative Abstinence

INTERVENTIONS:
Behavioral: Recent Ejaculation — Participants are instructed to ejaculate at least once within 36 hours prior to radical prostatectomy. This behavioral intervention is used to evaluate its effect on seminal vesicle volume and intraoperative dissection parameters.
  Other Names: Ejaculation within 36 hours before surgery
  Arms: Recent Ejaculation Group
Behavioral: Preoperative Abstinence — Participants are instructed to abstain from ejaculation for at least 72 hours prior to radical prostatectomy. This behavioral intervention is used to assess whether prolonged seminal vesicle filling affects intraoperative anatomy and dissection.
  Other Names: Ejaculatory Abstinence ≥72 hours
  Arms: Abstinence Group

SUMMARY:
The goal of this clinical trial is to learn if recent ejaculation or abstinence before surgery affects seminal vesicle size and dissection-related surgical factors in adult men with prostate cancer undergoing radical prostatectomy. The main questions it aims to answer are:

Does ejaculation within 36 hours before surgery reduce seminal vesicle size compared to abstinence of 72 hours or more?

Does seminal vesicle size affect the ease or difficulty of surgical dissection during radical prostatectomy?

Researchers will compare an ejaculation group to an abstinence group to see if seminal vesicle volume and intraoperative surgical parameters differ between them.

Participants will:

Follow specific instructions to either ejaculate or abstain before surgery

Undergo a transrectal ultrasound (TRUS) to measure seminal vesicle size after anesthesia but before surgery

Have their surgical dissection time and difficulty rated by the operating surgeon

DETAILED DESCRIPTION:
Radical prostatectomy (RP) remains a cornerstone treatment for localized prostate cancer. During RP, the anatomical dissection of seminal vesicles (SVs) can be challenging, and SV volume may influence intraoperative visibility, dissection ease, and the risk of complications.

Recent imaging studies suggest that ejaculatory activity significantly affects SV size. In particular, abstinence has been associated with larger SV volumes on MRI and TRUS, while ejaculation may lead to temporary SV shrinkage. These physiological changes, though well-documented radiologically, have not been systematically studied in a surgical setting.

This trial aims to explore whether ejaculatory behavior in the days before RP alters the surgical anatomy and impacts dissection-related metrics. Forty adult male patients with biopsy-confirmed prostate cancer, scheduled for RP, will be randomized in a 1:1 ratio into two groups:

Ejaculation group: At least one ejaculation within 36 hours preoperatively.

Abstinence group: No ejaculation for ≥72 hours before surgery.

Under anesthesia and prior to surgery, transrectal ultrasound (TRUS) will be performed to measure bilateral SV dimensions. The average volume will serve as the primary endpoint. Intraoperative outcomes include dissection time, visual clarity, and perceived difficulty rated by the primary surgeon using a Likert scale. SV volume from final pathology reports will also be collected and compared.

This is a low-risk, behavior-based interventional study involving no experimental drug or device. The main purpose is to assess whether preoperative sexual behavior can be optimized to improve surgical planning and efficiency. Alpha-blocker usage and other potential confounders will be documented and adjusted for in the analysis.

If significant anatomical or procedural differences are observed, findings from this study may inform future multicenter research and guide preoperative patient counseling for RP.

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged 18 years or older
* Histologically confirmed prostate cancer
* Scheduled for radical prostatectomy
* Able and willing to comply with assigned ejaculation or abstinence protocol
* Willing to complete preoperative questionnaire
* Willing to undergo transrectal ultrasound (TRUS) 12-14 hours before surgery
* Able to understand and sign informed consent

Exclusion Criteria:

* Prior bilateral seminal vesicle resection or congenital absence of seminal vesicles
* Anatomical abnormalities preventing SV identification
* Hormone therapy within 6 months before surgery
* Inability to recall ejaculation history in the past 3 days
* Inability to follow behavioral instructions or TRUS protocol
* Severe anorectal disease or history of anorectal surgery preventing TRUS
* Cognitive or psychiatric conditions impairing informed consent
* Incomplete data or poor-quality imaging
* Prior prostate cancer treatment
* Belonging to a vulnerable population (e.g., minors, prisoners, pregnant individuals, cognitively impaired, etc.)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-09 (Estimated)

PRIMARY OUTCOMES:
Seminal vesicle volume measured by preoperative transrectal ultrasound (TRUS) | 12-14 hours before surgery (afternoon prior to operation)
  Seminal vesicle volume is measured by the research investigator using transrectal ultrasound (TRUS) in the outpatient ultrasound room approximately 12-14 hours before surgery. Both vesicles are measured in three dimensions (length × width × height), and the average volume is calculated using the ellipsoid formula (L × W × H × 0.52). The values will be compared between groups with recent ejaculation versus abstinence.

SECONDARY OUTCOMES:
Dissection time of seminal vesicles during radical prostatectomy | During surgery (intraoperative)
  The time required for bilateral seminal vesicle dissection is recorded in minutes from surgical video or intraoperative notes.
Surgical difficulty score of seminal vesicle dissection | Immediately after SV dissection during surgery
  The primary surgeon rates the difficulty of SV dissection on a Likert scale from 1 (very easy) to 5 (very difficult), based on anatomical clarity and tissue handling.
Intraoperative visual clarity score of seminal vesicles | During SV dissection, intraoperatively
  The operating surgeon rates visual clarity of the surgical field (especially SV region) using a Likert scale from 1 (very poor) to 5 (excellent).
Seminal vesicle volume reported in postoperative pathology | Within 7 days after surgery (postoperative pathology report)
  Pathology reports include three-dimensional measurements of both SVs. Final volume is calculated using the same ellipsoid formula and compared with TRUS findings.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Cancer Center, Taipei, Outside U.S./Canada, Taiwan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional policies and IRB-approved protocols that limit data access to the research team. The dataset is small, single-center, and contains sensitive clinical and behavioral information. There is no current plan to develop a public repository or de-identified dataset for external use.

REFERENCES:
- [Background] Medved M, Sammet S, Yousuf A, Oto A. MR imaging of the prostate and adjacent anatomic structures before, during, and after ejaculation: qualitative and quantitative evaluation. Radiology. 2014 May;271(2):452-60. doi: 10.1148/radiol.14131374. Epub 2014 Feb 1. PMID 24495265
- [Background] Shin T, Kaji Y, Shukuya T, Nozaki M, Soh S, Okada H. Significant changes of T2 value in the peripheral zone and seminal vesicles after ejaculation. Eur Radiol. 2018 Mar;28(3):1009-1015. doi: 10.1007/s00330-017-5077-4. Epub 2017 Oct 6. PMID 28986624
- [Background] Yuruk E, Pastuszak AW, Suggs JM 3rd, Colakerol A, Serefoglu EC. The association between seminal vesicle size and duration of abstinence from ejaculation. Andrologia. 2017 Sep;49(7):10.1111/and.12707. doi: 10.1111/and.12707. Epub 2016 Sep 23. PMID 27660049